CLINICAL TRIAL: NCT02541383
Title: Study of Daratumumab in Combination With Bortezomib (VELCADE), Thalidomide, and Dexamethasone (VTD) in the First Line Treatment of Transplant Eligible Subjects With Newly Diagnosed Multiple Myeloma
Brief Title: A Study to Evaluate Daratumumab in Transplant Eligible Participants With Previously Untreated Multiple Myeloma
Acronym: Cassiopeia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone du Myelome (Network)
Collaborators: HOVON - Dutch Haemato-Oncology Association (Other); Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFM 2015-01; HO131 (Other: HOVON); 54767414MMY3006 (Other: J&J); 2014-004781-15 (EudraCT Number)
Record Dates: First submitted 2015-06-24; First posted 2015-09-04 (Estimated); Results first posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
Keywords: Untreated Multiple Myeloma; daratumumab
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Thalidomide; Dexamethasone; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A Part 1 (Other): Bortezomib (VELCADE), Thalidomide, and Dexamethasone (VTD)
  Interventions: Drug: Bortezomib (VELCADE), Thalidomide, and Dexamethasone (VTD)
- Arm B Part 1 (Experimental): Bortezomib (VELCADE), Thalidomide, and Dexamethasone (VTD) plus daratumumab
  Interventions: Drug: Bortezomib, Thalidomide, Dexamethasone (VTD) + daratumumab
- Arm A Part 2 (No Intervention): Observation
- Arm B Part 2 (Experimental): daratumumab
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Bortezomib (VELCADE), Thalidomide, and Dexamethasone (VTD) — Part 1: 4 Cycles of Bortezomib,Thalidomide and Dexamethasone induction therapy, followed by Autologous Stem Cell Transplantation, followed by 2 cycles of Bortezomib, Thalidomide and Dexamethasone consolidation
  Other Names: Arm A Part 1
  Arms: Arm A Part 1
Drug: Bortezomib, Thalidomide, Dexamethasone (VTD) + daratumumab — Part 1: 4 Cycles of Bortezomib, Thalidomide and Dexamethasone plus daratumumab 16mg/kg induction therapy, followed by Autologous Stem Cell Transplantation, followed by 2 cycles of Bortezomib, Thalidomide and Dexamethasone plus daratumumab 16 mg/kg consolidation
  Other Names: Arm B Part 1
  Arms: Arm B Part 1
Drug: Daratumumab — Daratumumab 16mg/kg every 8 weeks for 2 years
  Other Names: Arm B Part 2
  Arms: Arm B Part 2

SUMMARY:
The purpose of this study is to evaluate if the addition of daratumumab to Bortezomib, Thalidomide and Dexamethasone will increase the stringent complete response rate after consolidation therapy and increase the progression free survival after daratumumab maintenance therapy in transplant eligible participants with previously untreated Multiple Myeloma.

DETAILED DESCRIPTION:
This is a randomized, open-label (identity of assigned treatment will be known to participants and study staff), 2-arm (2 treatment groups), multicenter study of daratumumab in participants diagnosed with previously untreated Multiple Myeloma who are eligible for high dose chemotherapy and autologous stem cell transplantation (transplantation of own bone marrow). Participants will be randomized (assigned by chance) to one of 2 treatment groups to either receive daratumumab plus bortezomib, thalidomide and dexamethasone or bortezomib, thalidomide and dexamethasone for induction (before transplantation) and consolidation (after transplantation) treatment. All responders will then be re-randomized (assigned by chance) to one of 2 treatment groups to receive maintenance treatment with daratumumab only or observation (no treatment). The study will include a 28-Day Screening Phase, a Treatment Phase of 6 treatment cycles (each cycle is 4 weeks in duration for total period of 30 weeks), and a Follow up Phase of 2 years. The total duration for each participant in the study will be approximately 138 weeks. The end of the study will occur approximately 5 years after the last participant is randomized in the second phase of the study. Disease assessments will be performed every 4 weeks in the first phase of the study and then every 8 weeks in the second phase of the study. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of previously untreated multiple myeloma (MM)
* Have a confirmed diagnosis and eligible for high dose chemotherapy and autologous stem cell transplantation, and an Eastern Cooperative Oncology Group (ECOG) performance status score of 0,1 or 2

Exclusion Criteria:

* previous treatment for Multiple Myeloma
* Primary amyloidosis, Plasma Cell Leukemia or Smoldering Multiple Myeloma
* Prior or concurrent exposure to systemic therapy or SCT (Stem Cell Transplantation) for any plasma cell dyscrasia, with the exception of an emergency use of a short course (equivalent of dexamethasone 40 mg/day for a maximum 4 days) of corticosteroids before treatment, or received an investigational drug or used an invasive investigational medical device within 4 weeks before Cycle 1, Day 1
* history of malignancy (other than Multiple Myeloma) within 10 years before the date of randomization, except for the following if treated and not active: basal cell or nonmetastatic squamous cell carcinoma of the skin, cervical carcinoma in situ, ductal carcinoma in situ of breast, or International Federation of Gynecology and Obstetrics (FIGO) Stage 1 carcinoma of the cervix
* known chronic obstructive pulmonary disease (COPD) or moderate to severe asthma
* any concurrent medical or psychiatric condition or disease (eg, autoimmune disease, active systemic disease, myelodysplasia) that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1085 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Moreau, Pr, Principal Investigator — CHU Nantes, France
Locations (107):
- Belgium (13):
  - BE-Antwerp-ZNA Stuivenberg, Antwerp
  - AZ St Jan Brugge Oostende AV, Bruges
  - Institut Jules Bordet, Brussels
  - UCL Saint-Luc, Brussels
  - UZ Brussel, Brussels
  - GHDC, Charleroi
  - UZ Gent, Ghent
  - CH Jolimont, La Louvière
  - University Hospital Leuven, Leuven
  - Domaine Universitaire du Sart Tilman, Liège
  - AZ Delta, Roeselare
  - AZ Turnhout, Turnhout
  - UCL Mont-Godinne, Yvoir
- France (67):
  - CHU Amiens Sud, Amiens
  - CHRU-Hôpital du Bocage, Angers
  - Centre Hospitalier d'Argenteuil Victor Dupouy, Argenteuil
  - Centre Hospitalier H.Duffaut, Avignon
  - Centre hospitalier de la Côte Basque, Bayonne
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Avicenne, Bobigny
  - Polyclinique Bordeaux Nord Acquitaine, Bordeaux
  - Hôpital de Fleyriat, Bourg-en-Bresse
  - CHRU Brest - Hôpital A. Morvan, Brest
  - CHU Caen - Côte de Nacre, Caen
  - Clinique du Parc, Castelnau-le-Lez
  - CH René Dubos, Cergy-Pontoise
  - Hôpital Privé Sévigné, Cesson-Sévigné
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - CH Chambéry, Chambéry
  - Hôpital d'Instruction des Armées Percy, Clamart
  - CHU d'Estaing, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - CHRU Dijon - Hôpital des Enfants, Dijon
  - Centre Hospitalier Général, Dunkirk
  - CHRU Hôpital A. Michallon, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - CHV André Mignot - Université de Versailles, Le Chesnay
  - CH de Chartres - Hôpital Louis Pasteur, Le Coudray
  - Centre Hospitalier, Le Mans
  - Clinique Victor Hugo, Le Mans
  - CHRU Hôpital Claude Huriez, Lille
  - GH de l'Institut Catholique Saint Vincent, Lille
  - Centre Hospitalier Universitaire (CHU) de Limoges, Limoges
  - Hôpital du Scorff, Lorient
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CH Meaux, Meaux
  - Hôpital de Mercy (CHR Metz-Thionville), Metz
  - Hopital Saint Eloi - CHU Montpellier, Montpellier
  - Hôpital E. Muller, Mulhouse
  - Centre Catherine de Sienne, Nantes
  - CHRU Hôtel Dieu, Nantes
  - Clinique de l'Archet, Nice
  - CHU Carémeau, Nîmes
  - CH La Source, Orléans
  - CHU Hôpital Saint Antoine, Paris
  - Hôpital Cochin, Paris
  - Hôpital Necker, Paris
  - Hôpital Saint Louis, Paris
  - Institut Curie, Paris
  - La Pitié, Paris
  - CH Saint Jean, Perpignan
  - CHRU - Hôpital du Haut Lévêque - Centre François Magendie, Pessac
  - Centre Hospitalier de Perigueux, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers - Pôle régional de Cancérologie, Poitiers
  - Ch Annecy Genevois, Pringy
  - Hôpital Robert Debré, Reims
  - CHRU Hôpital de Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Yves Le Foll, Saint-Brieuc
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Hospitalier, Saint-Quentin
  - CHU Strasbourg, Strasbourg
  - Strasbourg Oncologie Médicale, Strasbourg
  - Pôle IUCT Oncopole CHU, Toulouse
  - CHRU Hôpital Bretonneau, Tours
  - CHRU Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - CHBA, Vannes
- Netherlands (27):
  - MC Alkmaar, Alkmaar
  - Meander MC, Amersfoort
  - AMC, Amsterdam
  - OLVG, Amsterdam
  - Vumc, Amsterdam
  - Ziekenhuis Rijnstate, Arnhem
  - Amphia Hospital Breda, Breda
  - RdGG, Delft
  - Deventer zkh, Deventer
  - Albert Schweitzer zkh, Dordrecht
  - Maxima MC, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - UMCG, Groningen
  - Atrium MC/Zuyderland MC, Heerlen
  - Tergooiziekenhuizen, location Hilversum, Hilversum
  - Spaarne Gasthuis, Hoofddorp
  - MC Leeuwarden, Leeuwarden
  - LUMC, Leiden
  - MUMC, Maastricht
  - Antonius zkh, Nieuwegein
  - Radboudumc, Nijmegen
  - Erasmus MC, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Haga zkh, The Hague
  - Elisabeth zkh, Tilburg
  - UMCU, Utrecht
  - Isala Klinieken, Zwolle

REFERENCES:
- [Result] Moreau P, Attal M, Hulin C, Arnulf B, Belhadj K, Benboubker L, Bene MC, Broijl A, Caillon H, Caillot D, Corre J, Delforge M, Dejoie T, Doyen C, Facon T, Sonntag C, Fontan J, Garderet L, Jie KS, Karlin L, Kuhnowski F, Lambert J, Leleu X, Lenain P, Macro M, Mathiot C, Orsini-Piocelle F, Perrot A, Stoppa AM, van de Donk NW, Wuilleme S, Zweegman S, Kolb B, Touzeau C, Roussel M, Tiab M, Marolleau JP, Meuleman N, Vekemans MC, Westerman M, Klein SK, Levin MD, Fermand JP, Escoffre-Barbe M, Eveillard JR, Garidi R, Ahmadi T, Zhuang S, Chiu C, Pei L, de Boer C, Smith E, Deraedt W, Kampfenkel T, Schecter J, Vermeulen J, Avet-Loiseau H, Sonneveld P. Bortezomib, thalidomide, and dexamethasone with or without daratumumab before and after autologous stem-cell transplantation for newly diagnosed multiple myeloma (CASSIOPEIA): a randomised, open-label, phase 3 study. Lancet. 2019 Jul 6;394(10192):29-38. doi: 10.1016/S0140-6736(19)31240-1. Epub 2019 Jun 3. PMID 31171419
- [Result] Moreau P, Hulin C, Perrot A, Arnulf B, Belhadj K, Benboubker L, Bene MC, Zweegman S, Caillon H, Caillot D, Corre J, Delforge M, Dejoie T, Doyen C, Facon T, Sonntag C, Fontan J, Mohty M, Jie KS, Karlin L, Kuhnowski F, Lambert J, Leleu X, Macro M, Orsini-Piocelle F, Roussel M, Stoppa AM, van de Donk NWCJ, Wuilleme S, Broijl A, Touzeau C, Tiab M, Marolleau JP, Meuleman N, Vekemans MC, Westerman M, Klein SK, Levin MD, Offner F, Escoffre-Barbe M, Eveillard JR, Garidi R, Ahmadi T, Krevvata M, Zhang K, de Boer C, Vara S, Kampfenkel T, Vanquickelberghe V, Vermeulen J, Avet-Loiseau H, Sonneveld P. Maintenance with daratumumab or observation following treatment with bortezomib, thalidomide, and dexamethasone with or without daratumumab and autologous stem-cell transplant in patients with newly diagnosed multiple myeloma (CASSIOPEIA): an open-label, randomised, phase 3 trial. Lancet Oncol. 2021 Oct;22(10):1378-1390. doi: 10.1016/S1470-2045(21)00428-9. Epub 2021 Sep 13. PMID 34529931
- [Result] Moreau P, Hulin C, Perrot A, Arnulf B, Belhadj K, Benboubker L, Zweegman S, Caillon H, Caillot D, Avet-Loiseau H, Delforge M, Dejoie T, Facon T, Sonntag C, Fontan J, Mohty M, Jie KS, Karlin L, Kuhnowski F, Lambert J, Leleu X, Macro M, Orsini-Piocelle F, Roussel M, Schiano de Colella JM, van de Donk NW, Wuilleme S, Broijl A, Touzeau C, Tiab M, Marolleau JP, Meuleman N, Vekemans MC, Westerman M, Klein SK, Levin MD, Offner F, Escoffre-Barbe M, Eveillard JR, Garidi R, Hua W, Wang J, Tuozzo A, de Boer C, Rowe M, Vanquickelberghe V, Carson R, Vermeulen J, Corre J, Sonneveld P; Intergroupe Francophone du Myelome, the Dutch-Belgian Cooperative Trial Group for Hematology Oncology and the CASSIOPEIA Investigators. Bortezomib, thalidomide, and dexamethasone with or without daratumumab and followed by daratumumab maintenance or observation in transplant-eligible newly diagnosed multiple myeloma: long-term follow-up of the CASSIOPEIA randomised controlled phase 3 trial. Lancet Oncol. 2024 Aug;25(8):1003-1014. doi: 10.1016/S1470-2045(24)00282-1. Epub 2024 Jun 15. PMID 38889735
- [Derived] Kraeber-Bodere F, Jamet B, Zweegman S, Perrot A, Hulin C, Caillot D, Facon T, Leleu X, Belhadj K, Itti E, Karlin L, Bailly C, Levin MD, Minnema MC, Bodet-Milin C, de Keizer B, Corre J, Sonneveld P, Moreau P, Carlier T, Touzeau C. Prognostic value of premaintenance FDG PET/CT response in patients with newly diagnosed myeloma from the CASSIOPEIA trial. Blood. 2025 Dec 18;146(25):3050-3058. doi: 10.1182/blood.2025030084. PMID 40991848
- [Derived] Corre J, Vincent L, Moreau P, Hebraud B, Hulin C, Bene MC, Broijl A, Caillot D, Delforge M, Dejoie T, Facon T, Lambert J, Leleu X, Macro M, Perrot A, Zweegman S, Filleron T, Cabarrou B, van de Donk NWCJ, Maheo S, Hua W, Wang J, Krevvata M, Vanquickelberghe V, de Boer C, Tuozzo A, Borgsten F, Rowe M, Carson R, Wuilleme S, Sonneveld P. Daratumumab-bortezomib-thalidomide-dexamethasone for newly diagnosed myeloma: CASSIOPEIA minimal residual disease results. Blood. 2025 Aug 7;146(6):679-692. doi: 10.1182/blood.2024027620. PMID 40127397
- [Derived] Kraeber-Bodere F, Zweegman S, Perrot A, Hulin C, Caillot D, Facon T, Leleu X, Belhadj K, Itti E, Karlin L, Bailly C, Levin MD, Minnema MC, Jamet B, Bodet-Milin C, De Keizer B, Bene MC, Avet-Loiseau H, Sonneveld P, Pei L, Rigat F, De Boer C, Vermeulen J, Kampfenkel T, Lambert J, Moreau P. Prognostic value of positron emission tomography/computed tomography in transplant-eligible newly diagnosed multiple myeloma patients from CASSIOPEIA: the CASSIOPET study. Haematologica. 2023 Feb 1;108(2):621-626. doi: 10.3324/haematol.2021.280051. No abstract available. PMID 36263839
- [Derived] Alberge JB, Kraeber-Bodere F, Jamet B, Touzeau C, Caillon H, Wuilleme S, Bene MC, Kampfenkel T, Sonneveld P, van Duin M, Avet-Loiseau H, Corre J, Magrangeas F, Carlier T, Bodet-Milin C, Cherel M, Moreau P, Minvielle S, Bailly C. Molecular Signature of 18F-FDG PET Biomarkers in Newly Diagnosed Multiple Myeloma Patients: A Genome-Wide Transcriptome Analysis from the CASSIOPET Study. J Nucl Med. 2022 Jul;63(7):1008-1013. doi: 10.2967/jnumed.121.262884. Epub 2022 Jan 27. PMID 35086897
- [Derived] Hulin C, Offner F, Moreau P, Roussel M, Belhadj K, Benboubker L, Caillot D, Facon T, Garderet L, Kuhnowski F, Stoppa AM, Kolb B, Tiab M, Jie KS, Westerman M, Lambert J, Pei L, Vanquickelberghe V, De Boer C, Vermeulen J, Kampfenkel T, Sonneveld P, Van de Donk NWCJ. Stem cell yield and transplantation in transplant-eligible newly diagnosed multiple myeloma patients receiving daratumumab + bortezomib/thalidomide/dexamethasone in the phase 3 CASSIOPEIA study. Haematologica. 2021 Aug 1;106(8):2257-2260. doi: 10.3324/haematol.2020.261842. No abstract available. PMID 33657786
- [Derived] Roussel M, Moreau P, Hebraud B, Laribi K, Jaccard A, Dib M, Slama B, Dorvaux V, Royer B, Frenzel L, Zweegman S, Klein SK, Broijl A, Jie KS, Wang J, Vanquickelberghe V, de Boer C, Kampfenkel T, Gries KS, Fastenau J, Sonneveld P. Bortezomib, thalidomide, and dexamethasone with or without daratumumab for transplantation-eligible patients with newly diagnosed multiple myeloma (CASSIOPEIA): health-related quality of life outcomes of a randomised, open-label, phase 3 trial. Lancet Haematol. 2020 Dec;7(12):e874-e883. doi: 10.1016/S2352-3026(20)30356-2. PMID 33242444
- See also: FDA approval — https://www.fda.gov/drugs/resources-information-approved-drugs/fda-approves-daratumumab-transplant-eligible-multiple-myeloma

RESULTS

PARTICIPANT FLOW:
Groups:
- VTd Only: All patients randomized to the VTd group (Bortezomib (VELCADE), Thalidomide, and Dexamethasone) at rando 1 (even those who didn't receive any study treatment), not re-randomized in maintenance phase.
- DVTd Only * Arm/Group Title: Characters Remaining: 91: All patients randomized to the DVTd group (Daratumumab, Bortezomib (VELCADE), Thalidomide, and Dexamethasone) at rando 1 (even those who didn't receive any study treatment), not re-randomized in maintenance phase.
- VTd-OBS: All patients randomized to the VTd group (Bortezomib (VELCADE), Thalidomide, and Dexamethasone) at rando 1 (even those who didn't receive any study treatment), re-randomized to observation
- VTd-DARA: All patients randomized to the VTd group (Bortezomib (VELCADE), Thalidomide, and Dexamethasone) at rando 1 (even those who didn't receive any study treatment), re-randomized to daratumumab monotherapy
- DVTd-OBS: All patients randomized to the DVTd group (Daratumumab, Bortezomib (VELCADE), Thalidomide, and Dexamethasone) at rando 1 (even those who didn't receive any study treatment), re-randomized to observation.
- DVTd-DARA: All patients randomized to the DVTd group (Daratumumab, Bortezomib (VELCADE), Thalidomide, and Dexamethasone) at rando 1 (even those who didn't receive any study treatment), re-randomized to daratumumab monotherapy.
Period: Overall Study
Arm/Group | VTd Only | DVTd Only * Arm/Group Title: Characters Remaining: 91 | VTd-OBS | VTd-DARA | DVTd-OBS | DVTd-DARA
Started | 114 | 85 | 215 | 213 | 229 | 229
Completed | 53 | 38 | 165 | 170 | 205 | 204
Not Completed | 61 | 47 | 50 | 43 | 24 | 25
Not completed — Death | 50 | 37 | 48 | 41 | 21 | 25
Not completed — Lost to Follow-up | 5 | 3 | 1 | 1 | 3 | 0
Not completed — Consent withdrawn | 5 | 6 | 1 | 1 | 0 | 0
Not completed — Sponsor's decision | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- VTd Only: Bortezomib (VELCADE), Thalidomide, and Dexamethasone (VTD), not re-randomized in maintenance phase
- DVTd Only: Daratumumab in combination with Bortezomib (VELCADE), Thalidomide, and Dexamethasone (VTD), not re-randomized in maintenance phase
- VTd-OBS: Bortezomib (VELCADE), Thalidomide, and Dexamethasone (VTD) re-randomized to observation
- VTd-DARA: Bortezomib (VELCADE), Thalidomide, and Dexamethasone (VTD) re-randomized to daratumumab monotherapy
- DVTd-OBS: Daratumumab in combination with Bortezomib (VELCADE), Thalidomide, and Dexamethasone (VTD) re-randomized to observation
- DVTd-DARA: Daratumumab in combination with Bortezomib (VELCADE), Thalidomide, and Dexamethasone (VTD) re-randomized to daratumumab monotherapy
- Total: Total of all reporting groups
Arm/Group | VTd Only | DVTd Only | VTd-OBS | VTd-DARA | DVTd-OBS | DVTd-DARA | Total
Number analyzed (Participants) | 114 | 85 | 215 | 213 | 229 | 229 | 1085
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (6.36) | 57.8 (7.5) | 56 (6.96) | 56.3 (7.38) | 56.8 (6.83) | 56.4 (6.79) | 56.6 (6.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 37 | 94 | 87 | 96 | 94 | 450
  Male | 72 | 48 | 121 | 126 | 133 | 135 | 635
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  BELGIUM | 15 | 5 | 11 | 18 | 23 | 17 | 89
  FRANCE | 70 | 64 | 191 | 169 | 177 | 183 | 854
  NETHERLANDS | 29 | 16 | 13 | 26 | 29 | 29 | 142
Baseline ISS Stage [Number; unit: participants] — The International Staging System (ISS) for Multiple Myeloma was established by the International Myeloma Working Group (IMWG) in 2005. Sβ2M = Serum β2 microglobulin.
  Stage I is defined by Sβ2M < 3.5 mg/L and serum albumin ≥ 3.5 g/dL - Stage II is defined by Sβ2M < 3.5 mg/L and serum albumin < 3.5 g/dL; or β2M ≥ 3.5 mg/L and < 5.5 mg/L, irrespective of serum albumin - Stage III is defined by Sβ2M ≥ 5.5 mg/L Stage I is considered to have a better prognosis and stage III a worse prognosis.
  participants
    I | 47 | 25 | 88 | 93 | 83 | 96 | 432
    II | 52 | 41 | 96 | 85 | 118 | 96 | 488
    III | 15 | 19 | 31 | 35 | 28 | 37 | 165
Baseline Type of Myeloma [Number; unit: participants] — Multiple myeloma has different types of monoclonal proteins. These types are based on the immunoglobulin (protein) produced by the myeloma cell and they are identified by immunofixation method. The five types of heavy protein chains are G, A, D, E, and M.
  The two types of light protein chains are kappa (κ) and lambda (λ). The myeloma cells may secrete heavy and light protein chains (i.e. IgG Kappa) but also only light protein chains.
  Row "Biclonal" = the myeloma cells (plasmocytes) produce two immunoglobulins with heavy chains - Row "negative immunofixation" = absence of monoclonal proteins
  participants
    Biclonal | 1 | 2 | 10 | 8 | 5 | 5 | 31
    IgA | 15 | 14 | 46 | 43 | 36 | 37 | 191
    IgD | 3 | 1 | 3 | 7 | 2 | 2 | 18
    IgG | 79 | 54 | 126 | 128 | 159 | 138 | 684
    IgM | 0 | 0 | 1 | 1 | 0 | 1 | 3
    Kappa | 11 | 9 | 17 | 18 | 17 | 27 | 99
    Lambda | 3 | 5 | 10 | 7 | 8 | 17 | 50
    Negative immunofixation | 2 | 0 | 2 | 1 | 2 | 2 | 9
Time since initial diagnosis to randomization (months) [Mean (Standard Deviation); unit: months] | 1.6 (2.65) | 1.3 (0.96) | 1.2 (0.86) | 1.2 (0.87) | 1.2 (1.08) | 1.2 (0.95) | 1.2 (1.25)
Presence of diffuse myeloma-related osteopenia [Number; unit: participants]
  No | 100 | 76 | 197 | 194 | 203 | 208 | 978
  Yes | 14 | 9 | 18 | 17 | 25 | 19 | 102
  Missing | 0 | 0 | 0 | 2 | 1 | 2 | 5
Presence of evaluable bone marrow assessment [Number; unit: participants]
  No | 3 | 0 | 3 | 3 | 4 | 6 | 19
  Yes | 111 | 85 | 212 | 210 | 225 | 223 | 1066
Bone marrow cellularity [Number; unit: participants] — A sample of bone marrow aspirate was analyzed to count the cells and assess the cellular richness
  participants
    Hypercellular | 30 | 28 | 62 | 63 | 62 | 46 | 291
    Indeterminate | 1 | 3 | 8 | 8 | 6 | 8 | 34
    Moderately cellular | 24 | 19 | 50 | 42 | 41 | 47 | 223
    Normocellular | 52 | 31 | 78 | 93 | 101 | 112 | 467
    Severely acellular | 5 | 3 | 13 | 5 | 14 | 10 | 50
    Missing | 2 | 1 | 4 | 2 | 5 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Post-Consolidation Stringent Complete Response (sCR) Rate
Description: Post-consolidation sCR rate is defined as the percentage of ITT subjects who achieved or maintained sCR status within 30 days of Day 100 post Autologous Stem Cell Transplant (ASCT). The sCR status is assessed using the computerized algorithm according to IMWG response criteria, and must be achieved on or prior to start of subsequent therapies. Subjects must not die or progress by Day 100 post ASCT.
  According to the IMWG consensus recommendations for multiple myeloma treatment response criteria from 2006, the stringent complete response (sCR) was defined by a negative immunofixation on the serum and urine, and a disappearance of any soft tissue plasmacytomas, and < 5% plasma cells in bone marrow, plus normal free-light chain ratio and the absence of clonal bone marrow plasma cells by immunohistochemistry, immunofluorescence or 2- to 4-color flow cytometry.
Time Frame: At day 100 post Autologous Stem Cell Transplant (ASCT), up to 114 days post ASCT
Population: All participants randomized in the first randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Part 1 | Arm B Part 1
Number analyzed (Participants) | 542 | 543
Participants | 110 | 157
Statistical Analysis 1: Comparison: Arm A Part 1 vs Arm B Part 1; Test type: Superiority; p = 0.0010, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.6, 95% CI 2-sided [1.21 to 2.12]

2. Primary Outcome: Progression Free Survival (PFS) Post Completion of Maintenance Therapy
Description: Progression Free Survival (PFS) post completion of maintenance therapy is defined as the duration from the date of second randomization to either progressive disease (according to the IMWG criteria specified in the protocol), or death, whichever occurs first (=all these considered as events) at the completion of Maintenance therapy.
Time Frame: From the date of second randomization to either progressive disease or death which ever occurred first, with a median follow-up time of 35.4 months (cut-off for analysis was 26 months after the last rando 2 date).
Population: All participants randomized in the second randomization even if they did not receive any study treatment dose.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm A Part 2: All patients randomized to the Observation group at rando 2 (whatever the treatment allocated at rando 1)
- Arm B Part 2: All patients randomized to the Daratumumab group at rando 2 even those who didn't receive any treatment dose (whatever the treatment allocated at rando 1).
  Daratumumab: Daratumumab 16mg/kg every 8 weeks for 2 years
Arm/Group | Arm A Part 2 | Arm B Part 2
Number analyzed (Participants) | 444 | 442
Months | 46.7 [40.0 to NA] — The upper limit of the Confidence Interval is not estimable due to insufficient number of participants with events. | NA [NA to NA] — The Median time to progression was not reached in this arm. Consequently, the lower and upper limit of the Confidence Interval is not available due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Arm A Part 2 vs Arm B Part 2; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.42 to 0.68]

3. Secondary Outcome: Progression Free Survival (PFS) From First Randomization up to the End of the Study
Description: Progression Free Survival (PFS) is defined as the duration from the date of first randomization to either progressive disease (according to the IMWG criteria specified in the protocol), or death, whichever occurs first (=all these considered as events) at the end of the study
Time Frame: From the date of first randomization to either progressive disease or death which ever occurred first, with a median follow-up time of 80.1 months at the end of the study
Population: All participants randomized in the first randomization even if they did not receive any study treatment dose.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm A - Part 1 up to End of Study: All patients randomized to the VTd group (Bortezomib (VELCADE), Thalidomide, and Dexamethasone) at rando 1 (whether they subsequently had rando 2 or not) even those who didn't receive any treatment dose.
- Arm B - Part 1 up to End of Study: All patients randomized to the DVTd group (Daratumumab in combination with Bortezomib (VELCADE), Thalidomide, and Dexamethasone) at rando 1 (whether they subsequently had rando 2 or not) even those who didn't receive any treatment dose.
Arm/Group | Arm A - Part 1 up to End of Study | Arm B - Part 1 up to End of Study
Number analyzed (Participants) | 542 | 543
Months | 52.8 [47.5 to 58.7] | 83.7 [70.2 to NA] — The upper limit of the Confidence Interval is not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Arm A - Part 1 up to End of Study vs Arm B - Part 1 up to End of Study; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.52 to 0.72]

ADVERSE EVENTS:
Time Frame: AEs that started during the treatment until 30 days after the last dose of study treatment, approximately 59 months, except for secondary malignancies and deaths followed until the end of the study.
Description: VTd & DVTd (Part 1) arms contain the SAEs/AEs considered treatment emergent (TEAE) to Part 1 only from the 1st dose and before 2nd rando or subsequent therapy (ST), or after 2nd rando if TEAE related to the Part 1 treatment.
  VTd-DARA & DVTd-DARA (Part 2) arms include SAEs/AEs considered TEAE to Part 2, from the 2nd rando up to 30 days after the last dose prior to ST.
  VTd-OBS & DVTd-OBS (Part 2) include SAEs/AEs from 2nd rando until 2 years + 30 days but prior to study discontinuation or ST.
Groups:
- VTd - Part 1: All patients randomized to the VTd group (Bortezomib (VELCADE), Thalidomide, and Dexamethasone) at rando 1 (whether they subsequently had rando 2 or not) and who received at least one dose of treatment.
  It includes deaths that occurred from the 1st randomization to the end of the study.
  For the all-cause mortality report, the at risk population also includes the patients randomized but who didn't receive any treatment.
- DVTd - Part 1: All patients randomized to the DVTd group (Daratumumab in combination with Bortezomib (VELCADE), Thalidomide, and Dexamethasone) at rando 1 (whether they subsequently had rando 2 or not) and who received at least one dose of treatment.
  It includes deaths that occurred from the 1st randomization to the end of the study.
  For the all-cause mortality report, the at risk population also includes the patients randomized but who didn't receive any treatment.
- VTd-OBS - Part 2: All patients randomized to the VTd group (Bortezomib (VELCADE), Thalidomide, and Dexamethasone) at rando 1 and to observation group (OBS) at rando 2.
  It includes deaths that occurred from the 2nd randomization to the end of the study.
  That means that all deaths reported in this arm are also reported in the arm VTd - Part 1.
- VTd-DARA - Part 2: All patients randomized to the VTd group (Bortezomib (VELCADE), Thalidomide, and Dexamethasone) at rando 1 and to daratumumab group (DARA) at rando 2 and who received at least one dose of treatment after Rando 2.
  It includes deaths that occurred from the 2nd randomization to the end of the study.
  That means that all deaths reported in this arm are also reported in the arm VTd - Part 1.
- DVTd-OBS - Part 2: All patients randomized to the DVTd group (Daratumumab in combination with Bortezomib (VELCADE), Thalidomide, and Dexamethasone) at rando 1 and to observation group (OBS) at rando 2.
  It includes deaths that occurred from the 2nd randomization to the end of the study.
  That means that all deaths reported in this arm are also reported in the arm DVTd - Part 1.
- DVTd-DARA - Part 2: All patients randomized to the DVTd group (Daratumumab in combination with Bortezomib (VELCADE), Thalidomide, and Dexamethasone) at rando 1 and to daratumumab group (DARA) at rando 2 and who received at least one dose of treatment after Rando 2.
  It includes deaths that occurred from the 2nd randomization to the end of the study.
  That means that all deaths reported in this arm are also reported in the arm DVTd - Part 1.
Arm/Group | VTd - Part 1 | DVTd - Part 1 | VTd-OBS - Part 2 | VTd-DARA - Part 2 | DVTd-OBS - Part 2 | DVTd-DARA - Part 2
All-Cause Mortality (participants affected / at risk) | 139/542 | 83/543 | 48/215 | 41/211 | 21/229 | 25/229
Serious Adverse Events (participants affected / at risk) | 261/538 | 264/536 | 35/215 | 58/211 | 50/229 | 43/229
Other Adverse Events (participants affected / at risk) | 529/538 | 534/536 | 170/215 | 194/211 | 198/229 | 205/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VTd - Part 1 (N=538) | DVTd - Part 1 (N=536) | VTd-OBS - Part 2 (N=215) | VTd-DARA - Part 2 (N=211) | DVTd-OBS - Part 2 (N=229) | DVTd-DARA - Part 2 (N=229)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 12 | 7 | 0 | 0 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 16 | 12 | 0 | 1 | 0 | 0
Haemolytic Uraemic Syndrome (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Histiocytosis Haematophagic (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 3 | 7 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 8 | 22 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 12 | 1 | 0 | 0 | 0
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arrhythmia Supraventricular (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 6 | 1 | 0 | 2 | 1 | 1
Atrial Flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Atrial Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular Block (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac Amyloidosis (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Cardiac Failure (Cardiac disorders) | 5 | 2 | 0 | 0 | 0 | 0
Cardiac Failure Acute (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Coronary Artery Stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mitral Valve Prolapse (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Paroxysmal Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ventricular Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fanconi Syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Diverticular Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Duodenal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hernial Eventration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Inflammatory Bowel Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 6 | 0 | 1 | 0 | 1
Neutropenic Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic Cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 4 | 0 | 0 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 6 | 0 | 2 | 0 | 0
Asthenia (General disorders) | 3 | 3 | 0 | 0 | 1 | 0
Chest Discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 3 | 2 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
General Physical Health Deterioration (General disorders) | 3 | 6 | 1 | 0 | 0 | 0
Hernia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperthermia (General disorders) | 2 | 3 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Influenza Like Illness (General disorders) | 1 | 0 | 0 | 1 | 1 | 0
Malaise (General disorders) | 1 | 2 | 0 | 0 | 1 | 0
Medical Device Site Joint Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mucosal Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 22 | 15 | 0 | 0 | 0 | 2
Sudden Death (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatocellular Injury (Hepatobiliary disorders) | 0 | 3 | 0 | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anaphylactic Shock (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 2 | 1 | 0 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anal Abscess (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bacterial Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bacterial Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Bartholinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 7 | 0 | 2 | 1 | 1
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis Staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Chronic Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Clostridial Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Clostridium Colitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Clostridium Difficile Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cytomegalovirus Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cytomegalovirus Infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Cytomegalovirus Oesophagitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Dermo-Hypodermitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Device Related Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Eczema Infected (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Endocarditis Staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Enterococcal Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Epstein-Barr Virus Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Escherichia Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Escherichia Sepsis (Infections and infestations) | 3 | 2 | 0 | 0 | 0 | 0
Fungal Oesophagitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Gastroenteritis Salmonella (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpes Zoster Meningitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infectious Colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infective Thrombosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 4 | 0 | 1 | 0 | 0
Intervertebral Discitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Intestinal Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Legionella Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lower Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 2 | 5 | 3 | 3 | 4 | 3
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Metapneumovirus Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Pneumococcal Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumocystis Jirovecii Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 4 | 0 | 1 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 9 | 21 | 2 | 4 | 4 | 7
Pneumonia Acinetobacter (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia Bacterial (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Pneumonia Escherichia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia Fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia Haemophilus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia Influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia Legionella (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia Parainfluenzae Viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia Pneumococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia Pseudomonal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0
Pneumonia Viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Salmonella Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 11 | 7 | 1 | 0 | 0 | 1
Septic Shock (Infections and infestations) | 2 | 4 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Skin Bacterial Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Spinal Cord Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal Sepsis (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 0
Streptococcal Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Streptococcal Endocarditis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Streptococcal Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Streptococcal Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Systemic Mycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Thrombophlebitis Septic (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Varicella Zoster Virus Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0
Viral Diarrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral Infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0
Viral Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Blood Stem Cell Harvest Failure (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 0 | 0
Burns Second Degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fractured Sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0
Jaw Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Perirenal Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Product Preparation Error (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 5 | 3 | 0 | 1 | 0 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 3 | 2 | 1 | 0 | 0 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 0 | 0 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
General Physical Condition Abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic Enzyme Abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Cell Death (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 4 | 0 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 3 | 3 | 0 | 0 | 0 | 0
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fluid Overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fluid Retention (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 9 | 0 | 0 | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 0 | 0 | 0
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Compression (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 1 | 1 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Anaplastic Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2 | 2 | 0 | 2
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Blastic Plasmacytoid Dendritic Cell Neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Gastrointestinal Tract Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0
Lip Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 1 | 0
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Natural Killer-Cell Lymphoblastic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 2 | 1 | 1
Renal Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1 | 2 | 0 | 1
T-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Acute Motor-Sensory Axonal Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Amnestic Disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Autonomic Neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebellar Haematoma (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cervicobrachial Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Epidural Lipomatosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hemiparaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 2 | 2 | 1 | 0 | 0 | 0
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 16 | 11 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 4 | 1 | 0 | 0 | 0 | 0
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 2 | 0 | 1 | 1 | 1 | 2
Seizure (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 5 | 1 | 0 | 0 | 0 | 0
Status Epilepticus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0
Transient Global Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 2 | 0 | 1 | 0 | 0
Device Breakage (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0
Abnormal Behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 0 | 1 | 0
Anxiety Disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0
Delusional Disorder, Unspecified Type (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 4 | 2 | 0 | 0 | 0 | 0
Major Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mental Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 3 | 3 | 0 | 1 | 0 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cystitis Haemorrhagic (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 0
Myeloma Cast Nephropathy (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 3 | 1 | 1 | 0 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal Tubular Necrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Genital Prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Uterine Cervical Metaplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 1 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 0 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Eosinophilic Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Idiopathic Interstitial Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 0 | 0 | 0 | 0
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 1 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 20 | 8 | 0 | 0 | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus Polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute Generalised Exanthematous Pustulosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug Reaction with Eosinophilia and Systemic Symptoms (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arteritis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 7 | 3 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 2 | 0 | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Peripheral Artery Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vena Cava Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Venous Thrombosis (Vascular disorders) | 1 | 2 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VTd - Part 1 (N=538) | DVTd - Part 1 (N=536) | VTd-OBS - Part 2 (N=215) | VTd-DARA - Part 2 (N=211) | DVTd-OBS - Part 2 (N=229) | DVTd-DARA - Part 2 (N=229)
Anaemia (Blood and lymphatic system disorders) | 78 | 74 | 7 | 8 | 4 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 13 | 27 | 1 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 16 | 30 | 1 | 1 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 65 | 106 | 5 | 14 | 12 | 19
Neutropenia (Blood and lymphatic system disorders) | 83 | 149 | 6 | 7 | 4 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 72 | 109 | 4 | 7 | 4 | 10
Vertigo (Ear and labyrinth disorders) | 43 | 40 | 6 | 5 | 5 | 6
Vision Blurred (Eye disorders) | 31 | 23 | 1 | 1 | 1 | 2
Abdominal Pain (Gastrointestinal disorders) | 22 | 36 | 4 | 7 | 4 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 28 | 31 | 5 | 5 | 5 | 8
Constipation (Gastrointestinal disorders) | 255 | 271 | 2 | 10 | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 92 | 105 | 10 | 33 | 16 | 25
Dry Mouth (Gastrointestinal disorders) | 20 | 27 | 2 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 129 | 159 | 2 | 33 | 4 | 10
Stomatitis (Gastrointestinal disorders) | 102 | 93 | 1 | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 50 | 83 | 2 | 31 | 3 | 8
Asthenia (General disorders) | 159 | 176 | 27 | 35 | 26 | 26
Chills (General disorders) | 22 | 47 | 1 | 8 | 1 | 0
Fatigue (General disorders) | 85 | 75 | 9 | 14 | 17 | 16
Influenza Like Illness (General disorders) | 30 | 34 | 20 | 21 | 29 | 32
Injection Site Erythema (General disorders) | 28 | 31 | 0 | 0 | 0 | 0
Malaise (General disorders) | 25 | 35 | 4 | 6 | 3 | 2
Oedema Peripheral (General disorders) | 154 | 166 | 8 | 9 | 9 | 13
Pyrexia (General disorders) | 104 | 133 | 7 | 20 | 17 | 18
Hypogammaglobulinaemia (Immune system disorders) | 29 | 48 | 7 | 30 | 9 | 30
Bronchitis (Infections and infestations) | 79 | 107 | 71 | 77 | 63 | 93
Gastroenteritis (Infections and infestations) | 5 | 15 | 13 | 16 | 16 | 22
Herpes Zoster (Infections and infestations) | 21 | 27 | 26 | 14 | 39 | 17
Nasopharyngitis (Infections and infestations) | 33 | 60 | 20 | 37 | 29 | 39
Pneumonia (Infections and infestations) | 18 | 19 | 6 | 7 | 8 | 12
Rhinitis (Infections and infestations) | 19 | 34 | 9 | 19 | 13 | 20
Sinusitis (Infections and infestations) | 17 | 20 | 15 | 18 | 9 | 13
Upper Respiratory Tract Infection (Infections and infestations) | 20 | 40 | 9 | 29 | 27 | 35
Weight Decreased (Investigations) | 39 | 38 | 1 | 3 | 3 | 4
Decreased Appetite (Metabolism and nutrition disorders) | 36 | 39 | 2 | 1 | 3 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 23 | 31 | 1 | 1 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 26 | 24 | 20 | 27 | 31
Back Pain (Musculoskeletal and connective tissue disorders) | 48 | 49 | 32 | 19 | 31 | 26
Bone Pain (Musculoskeletal and connective tissue disorders) | 82 | 68 | 18 | 24 | 14 | 19
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 38 | 33 | 10 | 15 | 3 | 9
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 9 | 17 | 6 | 8 | 16 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 34 | 40 | 7 | 11 | 8 | 20
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 44 | 36 | 3 | 9 | 11 | 17
Dizziness (Nervous system disorders) | 32 | 36 | 1 | 2 | 4 | 5
Dysgeusia (Nervous system disorders) | 34 | 50 | 1 | 1 | 1 | 1
Headache (Nervous system disorders) | 42 | 44 | 5 | 10 | 8 | 6
Paraesthesia (Nervous system disorders) | 114 | 127 | 4 | 21 | 10 | 15
Peripheral Sensory Neuropathy (Nervous system disorders) | 340 | 325 | 24 | 31 | 27 | 39
Tremor (Nervous system disorders) | 58 | 72 | 0 | 2 | 0 | 2
Anxiety (Psychiatric disorders) | 47 | 61 | 3 | 4 | 6 | 3
Insomnia (Psychiatric disorders) | 81 | 64 | 5 | 8 | 5 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 90 | 19 | 41 | 23 | 39
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 63 | 78 | 2 | 20 | 6 | 9
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 25 | 27 | 5 | 3 | 6 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 23 | 45 | 6 | 21 | 10 | 14
Dry Skin (Skin and subcutaneous tissue disorders) | 35 | 29 | 2 | 4 | 6 | 5
Eczema (Skin and subcutaneous tissue disorders) | 7 | 18 | 4 | 11 | 4 | 7
Erythema (Skin and subcutaneous tissue disorders) | 50 | 61 | 1 | 14 | 1 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 25 | 2 | 17 | 6 | 7
Rash (Skin and subcutaneous tissue disorders) | 64 | 80 | 4 | 17 | 7 | 8
Hypertension (Vascular disorders) | 30 | 51 | 4 | 18 | 13 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT02541383/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT02541383/SAP_001.pdf